CLINICAL TRIAL: NCT01551342
Title: Evaluation Of Zetiq's Novel Cell Detect Technology For Detection Of Bladder Cancer In Urine Cytology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zetiq Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: ZT-CL-04B
Record Dates: First submitted 2012-03-07; First posted 2012-03-12 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2013-08

CONDITIONS: Bladder Cancer Transitional Cell Carcinoma
Keywords: bladder cancer; Transitional cell carcinoma (TCC)
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cystoscopic surveillance, TURT or Cystectomy: The following subjects will be enrolled: Subjects previously diagnosed with bladder cancer undergoing routine cystoscopic surveillance, TURT or Cystectomy.

SUMMARY:
* This study includes two semi-consecutive parts:

  * Part I Open label, controlled, Calibration part aimed to calibrate the CellDetect® device for identifying bladder cancer cells in urine samples.
  * Part II Prospective, controlled, blinded part to determine the performance of the CellDetect® device in monitoring bladder cancer recurrence in patients with a history of TCC, using urine cytology samples
* The following subjects will be enrolled:

Subjects previously diagnosed with bladder cancer undergoing routine cystoscopic surveillance, TURT or Cystectomy.

DETAILED DESCRIPTION:
Study aim:

1. To calibrate the CellDetect® device for detecting TCC in urine cytology samples.
2. Determine the performance of the CellDetect® device in identifying TCC recurrence in patients with a history of TCC using urine cytology samples.

The study includes two parts:

Part I Open label, controlled, Calibration part aimed to calibrate the CellDetect® device for identifying bladder cancer cells in urine samples.

Part II Prospective, controlled, blinded part to determine the performance of the CellDetect® device in monitoring bladder cancer recurrence in in patients with a history of TCC, using urine cytology samples

* The following subjects will be enrolled: Subjects previously diagnosed with bladder cancer undergoing routine cystoscopic surveillance, TURT or Cystectomy.

Part I - up to 200 urine eligible samples Part II - up to 300 urine eligible samples

Endpoints:

1. To calibrate the CellDetect® device for identifying TCC in urine cytology samples.
2. To determine the performance of the CellDetect® device in identifying recurrence of TCC in urine samples.

ELIGIBILITY:
Part A:

*Inclusion Criteria Inclusion criteria will be different for each group subjects.

Group A (Monitoring group):

1. Subjects diagnosed with bladder cancer undergoing routine cystoscopic surveillance, who had normal cystoscopies for at least 12 months..
2. Ability to provide informed consent
3. Age > 18 years

Group B (Positive group):

1. Subject undergoing TURT or cystectomy due to any of the following reasons:

   * Subjects with suspected or known TCC (hematuria subjects)
   * Subjects with previously diagnosed TCC undergoing routine cystoscopic surveillance.
2. Ability to provide informed consent
3. Age > 18 years

Exclusion Criteria

1. Participation in another clinical trial within last 30 days.
2. Known pregnancy on day of screening.

Part B:

*Inclusion Criteria

Subjects meeting the following criteria (all of them) will be included in the study:

1. Subject with a documented history of TCC and who are undergoing routine cystoscopic surveillance, TURBT or cystectomy
2. At least 4 weeks have passed since any treatment for TCC (including cystoscopy and/or TURBT procedures)
3. Ability to provide informed consent
4. Age ≥ 18 years old

   * Exclusion Criteria

Subjects complying with any of the following exclusion criteria will be excluded from the study:

1. Subject with catheters, neobladder or kidney stones.
2. Subject unable to provide a spontaneous urine sample.
3. Subject currently under any cancer drug treatment.
4. No biopsy results available for subjects with positive findings on cystoscopy test, TURBT or cystectomy. [Note: such subjects will be excluded after recruitment and urine collection, as result of the delay in receiving biopsy results].
5. If more than 3 months have passed between urine sample collection and TURBT or cystectomy procedures, and no second sample was taken before undergoing TURBT, subject will be excluded from the study.
6. Subject undergoing TURBT or cystectomy whose biopsy results demonstrated abnormal findings other than TCC.
7. Subject participated in another clinical study within the last 30 days.
8. Known pregnancy on day of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The following subjects will be enrolled: Subjects previously diagnosed with bladder cancer undergoing routine cystoscopic surveillance, TURT or Cystectomy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-01

CONTACTS AND LOCATIONS:
Locations (7):
- Israel (7):
  - Emek Medical Center, Afula
  - Urology Department, Bnai Zion Medical Center, Haifa
  - Urology Department, Hadassah Medical Center Ein Kerem, Jerusalem
  - Urology Department, Meir Medical Center, Kfar Saba
  - Urology Department, Rabin Medical Center, Belinson Campus, Petah Tikva
  - Urology Department, Sourasky Medical Center, Tel Aviv
  - Urology Department, Sheba Medical Center, Tel Litwinsky